CLINICAL TRIAL: NCT04621045
Title: Feasibility and Preliminary Efficacy of a Novel YouTube Based Physical Activity Intervention in Overweight and Obese Adults at High Risk of Type 2 Diabetes
Brief Title: Active You: Feasibility of a Unique Physical Activity Program to Prevent Diabetes and Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jacob Kariuki, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19090134
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Risk Factor; Prediabetes; Overweight and Obesity; Sedentary Behavior
Keywords: Physical activity; Web-based; YouTube
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Sedentary Behavior; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: We will randomize 52 participants to either the PATH treatment group or wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Treatment Group (Experimental): The PATH group will be granted password protected access to one of the 3 PATH levels based on their baseline fitness status. The intervention is designed to help participants increase their baseline PA via health coaching, self-monitoring and pragmatic workout videos that provide convenient options for overcoming socio-environmental barriers to PA.
  Interventions: Behavioral: The Physical Activity for The Heart (PATH) intervention
- Wait-list control group (Active Comparator): Participants in this group will not have access to the PATH intervention until after 12 weeks when they cross over. After randomization, the control group will be provided with a copy of the Be Active Your Way booklet, developed by the Centers for Disease Control (CDC) to help individuals integrate PA in their daily lives.
  Interventions: Behavioral: Be Active Your Way Booklet

INTERVENTIONS:
Behavioral: The Physical Activity for The Heart (PATH) intervention — The web-based Physical Activity for The Heart (PATH) intervention leverages openly accessible platforms, such as YouTube, to proffer workout videos that match the participants preferences. Currently, PATH includes over 90 workout videos vetted by a team of experts and curated on the PATH website in 3 controlled levels of intensity (beginner, intermediate, proficient) to foster gradual progression from low to high intensity PA in accordance with the FITT-VP (frequency, intensity, time, type, volume, progression) principle.
  Arms: PATH Treatment Group
Behavioral: Be Active Your Way Booklet — Be Active Your Way booklet was developed by the Centers for Disease Control (CDC) to help individuals integrate PA in their daily lives. It simply encourages individuals to increase their PA gradually and gives them examples of things that they can do.
  Arms: Wait-list control group

SUMMARY:
Individuals who are overweight/obese are more vulnerable to type 2 diabetes (T2D). Current evidence suggests that PA, even without dietary prescription, can be efficacious in preventing T2D. Yet most Americans, especially those who are overweight/obese, are not physically active. Socioenvironmental barriers to physical activity (PA) such as body image concerns and limited access to fitness facilities contribute to the low levels of PA observed in overweight/obese adults. Web-based PA programs have been developed to address these barriers, but the outcomes have been marginal. Qualitative studies suggest that individuals who are overweight/obese prefer PA programs that feature people they can relate to especially in body size, fitness status and age. Previously, the investigators have included these preferences in a technology-based Physical Activity for The Heart (PATH) intervention that leverages open source platforms, such as YouTube, to promote PA in any setting. In this application, the investigators propose to test the feasibility and preliminary efficacy of PATH in promoting PA and reducing cardiometabolic risk in adults who are overweight/obese and at high risk of diabetes. In Aim 1 the investigators will conduct a 12-week randomized clinical trial including 52 adults who are overweight/obese and at high risk of diabetes to assess the feasibility and acceptability of PATH. In Aim 2 investigators will examine the trend in PA and cardiometabolic risk change from baseline to post-intervention. This approach is innovative because it leverages open source technologies to provide low-cost, action-oriented PA resources that match the preferences of adults who are overweight/obese. This contribution will be significant because PATH could offer a convenient, enjoyable and scalable program that features "similar others" to promote PA in overweight/obese adults at high risk of diabetes.

DETAILED DESCRIPTION:
Currently, only 20% of American adults attain the minimum 150 mins/week of MVPA recommended by the 2018 PA Guidelines for Americans. The low levels of PA are associated with the rising prevalence of obesity and T2D. Individuals who are overweight/obese need a higher volume of PA (~200-300 mins of weekly MVPA) to mitigate cardiometabolic risk, but they face complex multifaceted barriers that decrease their engagement in PA. Multiple studies exploring barriers and facilitators of PA among these individuals have emphasized the need for interventions that address weight-related impediments (e.g., stigma, fitness) and environmental barriers such as limited access to fitness facilities. In the last 2 decades web-based PA programs have been developed to address these barriers and to provide more interactive resources than those typically mailed to participants in home-based programs. In a recent analytic review of web-based PA interventions, 44 out of 72 studies reported significant increases in PA. However, 10 out of 13 studies focusing on adults who are overweight/obese reported no significant improvements in PA. Most of these studies employed interventions that are typically used in the general population (e.g., learning modules, email feedback, chat sessions) without adapting them to address barriers that are unique to individuals who are overweight/obese. Formative studies and social cognitive theory supports the need for PA interventions that feature individuals who are overweight/obese engaging in PA to motivate action and demonstrate success. In recent years, Internet ubiquity and creation of YouTube has enabled fitness experts across the globe to develop and share a wide variety of high quality workout videos designed to make PA convenient and enjoyable for all demographics. The investigators leveraged these resources and the aforementioned preference data to design an action-oriented PATH program tailored for individuals who are overweight/obese. The workout videos curated on PATH website were vetted by the study team and stakeholders. The investigators contribution in this project is expected to be a detailed understanding of how open sourced resources in interventions like PATH are received and utilized by overweight/obese adults.

ELIGIBILITY:
Inclusion Criteria:

1. 40-70 years old
2. BMI≥25
3. Have regular access to the internet (via computer or smart phone)
4. Less than 90 mins of self-reported moderate to vigorous physical activity per week
5. American Diabetes Association (ADA) risk ≥5
6. Available for pre and post-intervention assessments.

Exclusion Criteria:

1. Unstable conditions that may require supervised PA
2. Physical limitations that may prohibit engagement in MVPA
3. Pregnancy or intention to become pregnant during study, history of CVD
4. Current participation in a PA study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | At the end of study approximately 48 weeks after commencement of the study
  Will be indicated by ability to recruit, screen, and enroll the target sample within 6 months of commencing recruitment, and retention of ≥80% of the sample.
Feasibility of self-monitoring step count using wrist worn ActiGraph GT9X | At the end of study approximately 52 weeks after commencement of the study
  will be indicated by the proportion of the sample with ≥4days per week of valid Actigraph wear time (≥10hrs) during the entire course of the study.
Acceptability of PATH intervention | At the end of study approximately 52 weeks after commencement of the study
  Will be indicated by utilization data that will be collected via Web analytics, and a post-intervention survey will assess the intervention acceptability.

SECONDARY OUTCOMES:
Change from baseline in body mass index (BMI) at 12 weeks | Post-intervention at 12 weeks
  BMI will be measured using Fitbit Aria II scale provided to the participant by the study team. The study team will guide the participants on how to measure their BMI and will supervise the measurement via HIPAA compliant Zoom session.
Change from baseline in body fat percentage at 12 weeks | Post-intervention at 12 weeks
  Body fat percentage will be measured using Fitbit Aria II scale provided to the participant by the study team. The study team will guide the participants on how to measure their body fat and will supervise the measurement via HIPAA compliant Zoom session.
Change from baseline in waist circumference at 12 weeks | Post-intervention at 12 weeks
  Waist circumference will be measured using Perfect waist tape measure provided to the participant by the study team. The study team will guide the participants on how to take the measurement using a standard video and will be able to observe the outcome of the measurement via HIPAA compliant Zoom session.
Change from baseline in blood pressure (BP) at 12 weeks | Post-intervention at 12 weeks
  Both diastolic and systolic BP will be reported. The measurement will be done using automated OMRON BP machine provided to the participant by the study team. The study team will guide the participants on how to take blood pressure and will supervise the measurement via HIPAA compliant Zoom session.
Change from baseline in glycated hemoglobin (HbA1C) at 12 weeks | Post-intervention at 12 weeks
  The sample for HbA1C will be collected by participants at home using the dry blood spot method. The study team will guide the participants on how to take the sample using a standard video and will supervise the collection via HIPAA compliant Zoom session. The sample will be processed by CoreMedica lab using standard protocols
Change from baseline in lipids at 12 weeks | Post-intervention at 12 weeks
  The blood sample for lipids (LDL, HDL, and total cholesterol) will be collected by participants at home using the dry blood spot method. The study team will guide the participants on how to take the sample using a standard video and will supervise the collection via HIPAA compliant Zoom session. The sample will be processed by CoreMedica lab using standard protocols.
Change from baseline in the risk score for diabetes at 12 weeks | Post-intervention at 12 weeks
  The risk score for diabetes will be measured via the American Diabetes Association (ADA) Risk Calculator. The scores range from 0 to 10 with higher scores indicating high risk for developing type 2 diabetes.
Change from baseline in step count at 12 weeks | Post-intervention at 12 weeks
  Step count will be measured using a wrist worn ActiGraph GT9X link (about half the participants used Fitbit charge 2 due to device defects that we detected with Actigraph GT9X) during the entire study period. The study outcomes will focus on change from baseline to 12 weeks.
Change from baseline in light physical activity at 12 weeks | Post-intervention at 12 weeks
  Light physical activity will be measured using a waist worn ActiGraph GT3X accelerometer.
Change from baseline in moderate to vigorous physical activity (MVPA) at 12 weeks | Post-intervention at 12 weeks
  MVPA will be measured using a waist worn ActiGraph GT3X accelerometer.
Change from baseline in Barriers Exercise Self-efficacy (BARSE) scale at 12 weeks | Post-intervention at 12 weeks
  Participants will be asked to respond to the BARSE scale appraising their exercise self-efficacy. The scale range from 0 to 100, with higher scores indicating increased exercise self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kariuki, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Primay Health Network, Beaver Falls, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
t is our goal to make all data generated from this proposal available to other investigators without compromising the confidentiality of participants. Investigators who would like to do a secondary analysis of de-identified data can submit a formal request for the data including the proposal of their intended analysis to the PI at activeu@pitt.edu. The PI will review all requests and facilitate data access once approval is granted.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months after the end of the study
Access Criteria: Data access will be provided based on scientific merit of the proposed analysis, IRB approval and data agreement contract as deemed appropriate by University of Pittsburgh

REFERENCES:
- [Derived] Kariuki JK, Sereika S, Erickson K, Burke LE, Kriska A, Cheng J, Milton H, Hirshfield S, Ogutu D, Gibbs B. Feasibility and preliminary efficacy of a novel web-based physical activity intervention in adults with overweight/obesity: A pilot randomized controlled trial. Contemp Clin Trials. 2023 Oct;133:107318. doi: 10.1016/j.cct.2023.107318. Epub 2023 Aug 23. PMID 37625586

DOCUMENTS (1):
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04621045/ICF_000.pdf